CLINICAL TRIAL: NCT06496607
Title: A Phase 2, Randomized, Double-blind, Placebo-controlled, Multiple Dose-Ranging Study to Assess the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Solrikitug in Adult Participants With Asthma (RAINIER)
Brief Title: A Study to Evaluate Solriktug in Adult Participants With Asthma
Acronym: RAINIER
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Uniquity One (UNI) (Industry)
Collaborators: DevPro Biopharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NSI-8226-204
Record Dates: First submitted 2024-07-03; First posted 2024-07-11 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Solrikitug low dose subcutaneous injection (Experimental): Solrikitug
  Interventions: Biological: NSI-8226
- Solrikitug mid dose subcutaneous injection (Experimental): Solrikitug
  Interventions: Biological: NSI-8226
- Solrikitug high dose subcutaneous injection (Experimental): Solrikitug
  Interventions: Biological: NSI-8226
- Placebo subcutaneous injection (Placebo Comparator): Placebo
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: NSI-8226 — Solrikitug
  Arms: Solrikitug low dose subcutaneous injection
Biological: NSI-8226 — Solrikitug
  Arms: Solrikitug mid dose subcutaneous injection
Biological: NSI-8226 — Solrikitug
  Arms: Solrikitug high dose subcutaneous injection
Biological: Placebo — Placebo
  Arms: Placebo subcutaneous injection

SUMMARY:
Phase 2 study to evaluate the safety, tolerability, PK, immunogenicity, and pharmacodynamics of solriktug with adult participants with asthma.

DETAILED DESCRIPTION:
This is a 12-week randomized, double-blind, placebo-controlled Phase 2 clinical study to evaluate the safety, tolerability, PK, immunogenicity, and pharmacodynamics of 3 dose levels of solrikitug versus placebo on top of standard of care in adult participants with asthma.

Approximately 140 adult participants with asthma will be randomized. Participants will receive solrikitug, or placebo, administered via subcutaneous injection at the study site, over a 12-week treatment period. The study also includes a post-treatment follow-up period of 16 weeks.

ELIGIBILITY:
Key inclusion criteria:

* Participant must be aged 18 to 75 years of age.
* Documented diagnosis of asthma at least 12 months prior to Screening.
* Participants must be on maintenance asthma medications, for at least 3 months prior to screening: inhaled corticosteroid (ICS) in combination with long-acting beta agonist (LABA), or as part of an approved triple therapy for asthma (ICS/LABA/long-acting muscarinic antagonist [LAMA]).
* Participant has an ACQ-6 score ≥1.5 at Screening Visit.
* Participant has FEV1 of ≥50% to 90%, inclusive, of predicted normal value at Screening Visit 1.
* Evidence of asthma as documented by reversibility in FEV1 of ≥12% and ≥200 mL over the pre-salbutamol FEV1 at Screening Visit.

Key exclusion criteria:

* Female participant who is pregnant or breastfeeding.
* Participant is a current smoker, or former smoker with a smoking history of ≥10 pack-years.
* Participant has a known hypersensitivity to any component of the formulation of solrikitug, including any of the excipients, or a history of anaphylactic reaction to any therapeutic monoclonal antibody.
* Participant has history or evidence of any clinically significant cardiovascular, hematologic, hepatic, immunologic, metabolic, urologic, neurologic, dermatologic, psychiatric, renal and/or other major disease or malignancy, or any other condition (risks factors of pneumonia) that in the opinion of the Investigator might obfuscate the study data.
* Participant has an exacerbation of asthma requiring use of OCS or hospitalization in the 6 weeks prior to Screening or during the Screening Period.
* Participant has history or evidence of any clinically significant pulmonary condition, other than asthma.
* Lower respiratory tract infection within the 6 weeks prior to Screening.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2024-07-26 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
To assess the effect of multiple doses of solrikitug on blood eosinophil counts compared with placebo | Over weeks 8 and 12
  Change from baseline in blood eosinophil counts evaluated over Weeks 8 to 12

SECONDARY OUTCOMES:
To assess the safety and tolerability of multiple doses of solrikitug | To week 12
  Adverse events (AEs) and serious adverse events (SAEs)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew W Lee, MD, Study Director — Vice President, Clinical Research
Locations (61):
- United States (61):
  - Research Site 006, Mobile, Alabama
  - Research Site 076, Peoria, Arizona
  - Research Site 021, Huntington Beach, California
  - Research Site 082, La Mesa, California
  - Research Site 031, Los Angeles, California
  - Research Site 020, Newport Beach, California
  - Research Site 037, Rancho Cucamonga, California
  - Research Site 036, San Jose, California
  - Research Site 062, San Jose, California
  - Research Site 071, West Covina, California
  - Research Site 024, Englewood, Colorado
  - Research Site 001, Clearwater, Florida
  - Research Site 026, Cutler Bay, Florida
  - Research Site 069, DeLand, Florida
  - Research Site 025, Leesburg, Florida
  - Research Site 003, Miami, Florida
  - Research Site 030, Miami Gardens, Florida
  - Research Site 041, Tallahassee, Florida
  - Research Site 081, Tamarac, Florida
  - Research Site 080, Cordele, Georgia
  - Research Site 084, East Point, Georgia
  - Research Site 052, Savannah, Georgia
  - Research Site 065, Boise, Idaho
  - Research Site 022, Meridian, Idaho
  - Research Site 018, Winfield, Illinois
  - Research Site 019, Merrillville, Indiana
  - Research Site 011, Sioux City, Iowa
  - Research Site 005, Lafayette, Louisiana
  - Research Site 027, White Marsh, Maryland
  - Research Site 016, South Dartmouth, Massachusetts
  - Research Site 087, Dearborn, Michigan
  - Research Site 033, Farmington Hills, Michigan
  - Research Site 086, Southfield, Michigan
  - Research Site 032, Missoula, Montana
  - Research Site 014, Henderson, Nevada
  - Research Site 073, Queens Village, New York
  - Research Site 004, Gastonia, North Carolina
  - Research 013, Winston-Salem, North Carolina
  - Research Site 013, Winston-Salem, North Carolina
  - Research Site 075, Lima, Ohio
  - Research Site 061, Toledo, Ohio
  - Research Site 007, Edmond, Oklahoma
  - Research Site 009, Medford, Oregon
  - Research Site 045, Portland, Oregon
  - Research Site 083, DuBois, Pennsylvania
  - Research Site 063, Philadelphia, Pennsylvania
  - Research Site 046, Mauldin, South Carolina
  - Research Site 066, North Charleston, South Carolina
  - Research Site 038, Hendersonville, Tennessee
  - Research Site 028, Knoxville, Tennessee
  - Research Site 017, Boerne, Texas
  - Research Site 072, Brownsville, Texas
  - Research Site 085, Carrollton, Texas
  - Research Site 078, Conroe, Texas
  - Research Site 042, Dallas, Texas
  - Research Site 010, Dallas, Texas
  - Research Site 064, Frisco, Texas
  - Research Site 074, Greenville, Texas
  - Research Site 015, Houston, Texas
  - Research Site 010, McKinney, Texas
  - Research Site 023, Hampton, Virginia